CLINICAL TRIAL: NCT02211989
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses (0.5 mg to 200 mg) of BI 14332 CL as Powder in the Bottle Reconstituted With 0.1% Tartaric Acid Administered to Healthy Male Subjects. A Randomised and Placebo-controlled Trial, Double Blinded Within Dose Groups
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 14332 CL Powder in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1233.1
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BI 14332 CL (Experimental): single rising dose
  Interventions: Drug: BI 14332 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 14332 CL
  Arms: BI 14332 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability and pharmacokinetics, and pharmacodynamics of BI 14332 CL

ELIGIBILITY:
Inclusion Criteria:

* Healthy males were included based on a complete medical history, including the physical examination, vital signs (BP, HR), 12-lead ECG, and clinical laboratory tests
* Age ≥18 and Age ≤50 years
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, HR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which reasonably influenced the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range and of clinical relevance
* Inability to comply with the dietary regimen of the study centre
* Any ECG value outside the reference range and of clinical relevance including, but not limited to QRS interval >120 ms or a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms or QT >500 ms)
* A history of additional risk factors for Torsades des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* The use of concomitant medications that prolong the QT/QTc interval

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2006-02; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to day 16
Number of patients with clinically significant findings in vital signs (blood pressure, heart rate) | up to day 16
Number of patients with clinically significant findings ECG | up to day 16
Number of patients with clinically significant findings laboratory tests | up to day 16
Assessment of global tolerability by investigator on a 4-point scale | within 9 to 16 days after drug administration

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 192 hours after drug administration
tmax (time from dosing to maximum concentration) | up to 192 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 192 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 192 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 192 hours after drug administration
λz (terminal rate constant in plasma) | up to 192 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 192 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 192 hours after drug administration
CL/F (total clearance of the analyte in the plasma after extravascular administration) | up to 192 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 192 hours after drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | up to 120 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 120 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 120 hours after drug administration
Change in Dipeptidyl peptidase IV (DDP-IV) activity | up to 192 hours after drug administration